CLINICAL TRIAL: NCT03713827
Title: 24-Month Performance of a Glass-hybrid-restorative in Non-carious Cervical Lesions of Patients With Bruxism: A Split-mouth, Randomized Clinical Trial
Brief Title: Clinical Performance of a Glass Hybrid Restorative in NCCL's of Patients With Bruxism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ece Meral, principal investigator, Hacettepe University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KA-16020
Record Dates: First submitted 2018-10-15; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Bruxism; Noncarious Cervical Lesions
Keywords: glass hybrids; bruxism; Non carious cervical lesions
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Intervention Model Description: double blinded, split mouth, randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- "composite resin", "Ceram-x One Universal" (Active Comparator): tooth restoration with nano-ceramic composite resin "Ceram-x one Universal"
  Interventions: Device: tooth restoration
- "glass ionomer cement", "Equia Forte" (Active Comparator): Tooth restoration with glass ionomer cement (Glass hybrid restorative system) "Equia Forte"
  Interventions: Device: tooth restoration

INTERVENTIONS:
Device: tooth restoration — restoration of non carious cervical lesions with two different restorative materials

SUMMARY:
This is a double blinded, split mouth, randomized clinical study that evaluated the performance of a glass hybrid restorative material in non-carious servical lesions in patients with bruxism. The lesions were restored with glass hybrid restorative (Equia Forte) or nano ceramic composite resin (Ceram-x One). Restorations were evaluated after 24 months according to USPHS criteria and the data were evaluated.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the clinical performance of a glass-hybrid-restorative compared with a nano ceramic composite resin in non-carious cervical lesions (NCCLs) of patients with bruxism.

For this purpose, twenty-five patients having NCCLs and bruxism enrolled to the present study. Before treatment, the dimensions of the NCCLs were measured in depth, gingival-incisal height and mesio-distal width using a CPI probe. Degree of tooth wear (TWI) and gingival conditions (GI) are also recorded. A total of 148 NCCLs were randomly restored with a a glass-hybrid-restorative system (Equia Forte Fil, GC, Tokyo, Japan) or a nano ceramic composite resin (Ceram.X One Universal, Dentsply, DeTrey, Konstanz, Germany) and restorations were evaluated at baseline and after 6,12 and 24 months according to the modified-USPHS criteria. Data were analyzed with Chi- Square, Fisher's Exact Test, Mann Whitney-U and Cochran's Q tests (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* non-hospitalized, healthy patients that were seeking dental treatmen
* occlusally contacted teeth

Exclusion Criteria:

* Patients having intensive medical history
* Chronic periodontitis,
* high caries activity,
* extremely poor oral hygiene,
* teeth with restorations,
* mobility due to periodontal disease
* in contacted with removable prosthetic construction were excluded from the study

Ages: 42 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Retention Alpha for at least 90% of the restorations | 24 months
  The primary factor for determining the clinical performance of a restorative material is the retention rate. It represents the survival rates of the restorations after a period of time. According to ADA guidelines, a restorative material should show at leat 90% alpha retention rate after 18 months to be considered as clinically acceptable. The retention is assesed as alpha (retentive restoratation) or charlie (failed restoration). Clinical evaluation is performed to examine if the restoration is in place or has fallen.

SECONDARY OUTCOMES:
marginal adaptation score alpha | 24 months
  It represents the marginal integrity of the restorations. It is scored as alpha (perfect marginal adaptation), bravo (detectable marginal discrepency, clinically acceptable) or charlie (marginal crevice, clinically unacceptable). The examination of marginal adaptation is performed by clinical examination of the restoration with probe.

IPD SHARING:
Plan to Share IPD: Undecided